CLINICAL TRIAL: NCT06416644
Title: The PORTuguese Registry of Supera Supported Femoral-Fopliteal Revascularization (SupPORT Registry)
Acronym: SupPORT regist
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Divino Espírito Santo de Ponta Delgada (Other)
Responsible Party: Principal Investigator, Dr. Nelson Oliveira, Principal Investigator, Hospital do Divino Espírito Santo de Ponta Delgada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-HDES-2023-309
Record Dates: First submitted 2024-04-30; First posted 2024-05-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Lower Limb Ischemia; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Chronic Limb Ischemia; Atherosclerosis of Femoral Artery; Superficial Femoral Artery Stenosis; Superficial Femoral Artery Occlusion; Superficial Femoral Artery Disease; Superficial Femoral Artery Lesions; Popliteal Artery Occlusion; Popliteal Artery Stenosis; Popliteal Arterial Stenosis
Keywords: Supera; Vasculomimetic; Stent; Chronic limb-threatening ischemia; Chronic limb ischemia; Superficial femoral artery; popliteal artery
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supera implant (Experimental): Supera implant
  Interventions: Device: Supera Vasculomimetic Stent

INTERVENTIONS:
Device: Supera Vasculomimetic Stent — Femoral-popliteal revascularization with Supera Stent

SUMMARY:
The SupPORT Registry aims at collecting real-world from Portuguese centers performing femoral-popliteal revascularization with Supera (r) implants. This is a prospective non-randomized non-controlled consecutive registry.

DETAILED DESCRIPTION:
Primary endpoints (at hospitalization, 30 days, 6 months, 1 year)

1. Limb salvage
2. Target lesion revascularization (TLR)
3. Freedom from major adverse limb events (MALE - Major Amputation, any index limb revascularization)

Secondary endpoints (at hospitalization, 30 days, 6 months, 1 year)

1. Freedom from Major adverse cardiovascular events (5-point endpoint: Stroke, myocardial infarction/Acute coronary syndrome, Any limb revascularization, Decompensated Congestive Heart Failure, Cardiovascular death1)
2. All-cause death / Cardiovascular death
3. Primary Patency(defined by Duplex Ultrassound Scan [DUS]2) Primary-Assisted Patency, Secondary Patency
4. Ankle-Brachial Index (ABI)
5. Rutherford-Becker classification

Inclusion Criteria Clinical

* Evidence of symptomatic obstructive peripheral arterial disease
* Individuals aged 18 and older
* All-comer patients undergoing endovascular lower-limb revascularization with Supera® stent implantation in the superficial femoral (SFA) or popliteal arteries
* Patient or legal representative understand the SupPORT registry procedures, and have voluntarily provided informed written consent regarding their participation.
* Participant is willing to remain in the SupPORT Registry for at least 1 year.

Angiographic

* Target lesion is a primary atherosclerotic lesion or a restenosis occurring in a non-stented of the SFA or the popliteal artery, distancing at least ≥ 1 cm from any previously implanted vascular stent.
* Target lesion causes a ≥50% arterial obstruction (visually confirmed on digital subtraction angiography).

Exclusion criteria

* Any contraindication for peri-interventional or post-interventional anti-thrombotic therapy (including, but not restricted to Non-fractioned heparina, low-molecular weight heparina [LMWH], Clopidogrel, Ticagrelol, Ticlopidine, Acetylsalicylic acid, dipiridamol, direct thrombin [factor II] or factor Xa inhibitors, vitamin-K antagonists).
* Participation in other research study that may influence obtained results.
* Pregnant or breastfeeding women, or expected pregnancy to occur during the study period.
* Treatment of intrastent restenosis/occlusion of previous peripheral vascular stent.
* Non-corrected hemodynamically significant obstructive arterial disease of the ipsilateral inflow arteries (aorta, iliac arteries)

Procedure Protocol - Endovascular revascularization

• Participating centers are invited to maintain local practice standards, used in endovascular peripheral arterial revascularization. Pre-implant ballooning and peri-interventional anti-thrombotic therapy will be captured by the database. Intra-procedural and peri-procedural adjuncts are allowed, and will be recorded.

Follow-up Protocol

* Minimum follow-up will include a clinical assessment up to 30-days post-intervention, at 6 months, and at 1 year. Routine ABI is mandatory. Routine DUS is recommended.
* Post-interventional anti-thrombotic therapy will be captured by the database, and will follow international recommendations, but also local practice standards and will be at the discretion of the assisting-physician.

Data collection and storage

* Data will be inserted at each center by the Investigation team on an electronic platform, created and managed by Infortucano.
* Principal Investigators will have access to the enrolled center's participant data.
* System components

  1. Registry Database All data regarding each participant's records will be anonymously collected in a Central Database, where it will be stored. There are no limits to the number of participating centers.
  2. Web Application - SupPORT Registry

     1. Registry - The application will run on internet browser, with individual user authentication required for each Principal investigator. This application will allow the recording of the data and follow-up data by each participating center.
     2. Information extraction - Inserted data by each center/investigator will be only accessible to each center/investigator during the study period. The Registry administrator will have access privileges to all participants' data. The application will provide general tables/graphics with generic information throughout the study period, accessible to all investigators (number or participants per center, overall inclusion, to be defined). All inserted data will be exportable to CSV files, allowing import to Microsoft Excel or SPSS software.
     3. Technological architecture - All components are developed Microsoft.NET platform. The web application will be developed on ASP.NET 3.5/4.0. The Database Management System (DBMS) will be Microsoft SQL Server 2012/2019. The used Web Server will be Microsoft IIS 7.0.
     4. Storage - The Central System and DBMS will be lodged in Safe Cloud Microsoft Azure Servers (InforTucano). The application address will be www.rnsupport.com. Cloud Microsoft Azure Server Characteristics:
* Physical Location: Western Europe (The Netherlands)
* Data backups with differential archives of the previous 15 days
* Availability - 99,9 %
* Anti-virus ESET File Security for Windows Server
* Double-Firewall (Windows Server e Microsoft Azure Firewall)
* Test version: http://test.infortucano.pt/RegistoSupPORT

  * User: admin
  * Pwd: admin123

Statistical analysis Statistical analysis: Continuous variables with a normal distribution will be described as mean and standard deviation. Continuous variables are presented as median and interquartile range (IQR) if skewed and will be tested among groups using the Mann-Whitney U-Test for independent samples. Related variables will be compared with the Wilcoxon Signed Rank Test. Categorical variables will be presented as count and percentage and will be compared using the Pearson's χ2 test or the Fisher´s exact test in cases of low number of events. Life-table based analyses will be used for endpoint assessment. Kaplan-Meier curves will be created, and differences tested according to the log rank test. For association between baseline characteristics endpoints, a multivariable logistic regression model (including time as a co-variate) or a Cox hazards proportion model will be created including variables with α-value ≤0.10 on univariate analysis, if appropriate. Stepwise backward elimination of variables with a P-value >.050 will be also used during multivariable modelling. Confidence-intervals of 95% (95%CI) will be used and statistical significance will be considered for α<.05. All statistical analyses will be performed using Statistical Package for Social Sciences 21.0 (IBM Inc, Chicago, Ill, USA).

ELIGIBILITY:
Inclusion Criteria:

* Evidence of symptomatic obstructive peripheral arterial disease.
* All-comer patients undergoing endovascular lower-limb revascularization with Supera® stent implantation in the superficial femoral (SFA) or popliteal arteries.
* Patient or legal representative understand the SupPORT registry procedures, and have voluntarily provided informed written consent regarding their participation.
* Participant is willing to remain in the SupPORT Registry for at least 1 year.
* Target lesion is a primary atherosclerotic lesion or a restenosis occurring in a non-stented of the SFA or the popliteal artery, distancing at least ≥ 1 cm from any previously implanted vascular stent.
* Target lesion causes a ≥50% arterial obstruction (visually confirmed on digital subtraction angiography).

Exclusion Criteria:

* • Any contraindication for peri-interventional or post-interventional anti-thrombotic therapy (including, but not restricted to Non-fractioned heparina, low-molecular weight heparina [LMWH], Clopidogrel, Ticagrelol, Ticlopidine, Acetylsalicylic acid, dipiridamol, direct thrombin [factor II] or factor Xa inhibitors, vitamin-K antagonists).
* Participation in other research study that may influence obtained results.
* Pregnant or breastfeeding women, or expected pregnancy to occur during the study period.
* Treatment of intrastent restenosis/occlusion of previous peripheral vascular stent.
* Non-corrected hemodynamically significant obstructive arterial disease of the ipsilateral inflow arteries (aorta, iliac arteries)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from major limb amputation | 1 year
  Number of limbs surviving without above ankle amputation
Target Lesion Revascularization (TLR) | 1 year
  Number of target lesions requiring re-intervention
MALE - Major Adverse Limb Event | 1 year
  Composite endpoint Major Amputation, any index limb revascularization

SECONDARY OUTCOMES:
MACE - Major Adverse Cardiovascular Event | 1 year
  Composite 5-point endpoint: Stroke, myocardial infarction/Acute coronary syndrome, Any limb revascularization, Decompensated Congestive Heart Failure, Cardiovascular death
All-cause Death | 1 year
  Death from any cause
Cardiovascular-related death | 1 year
  Death from cardiovascular causes
Primary Patency, Primary Assisted Patency, Secondary Potency | 1 year
  Patency of target lesion, without any intervention, with additional interventions
Ankle-Brachial Index | 1 year
  Pressure index obtained from ankle and brachial arterial measurements
Rutherford-Becker Classification | 1 year

CONTACTS AND LOCATIONS:
Locations (15):
- Portugal (15):
  - Hospital de Faro - Centro Hospitalar do Algarve, Faro, Algarve
  - Hospital Divino Espírito Santo, Ponta Delgada, Azores
  - Hospital Garcia de Orta, Almada, Lisbon District
  - Centro Hospitalar Tâmega e Sousa, Penafiel, Porto District
  - Centro Hospitalar Vila Nova de Gaia e Espinho, Vila Nova de Gaia, Porto District
  - Hospital Santo Espírito Ilha Terceira, Angra do Heroísmo, Terceira
  - Centro Hospitalar Universitário de Coimbra, Coimbra
  - Hospital da Senhora da Oliveira de Guimarães, Guimarães
  - Hospital de Santa Marta - Centro Hospitalar Lisboa Central, Lisbon
  - Hospital Egas Moniz - Centro Hospitalar Lisboa Central, Lisbon
  - Hospital de Santa Maria - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar Universitário de Santo António, Porto
  - Centro Hospitalar São João, Porto
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, Vila Real
  - Centro Hospitalar Tondela Viseu, Viseu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao M, Hua Y, Zhao X, Jia L, Yang J, Liu B. Optimal Ultrasound Criteria for Grading Stenosis of the Superficial Femoral Artery. Ultrasound Med Biol. 2018 Feb;44(2):350-358. doi: 10.1016/j.ultrasmedbio.2017.10.001. Epub 2017 Nov 14. PMID 29150366
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334
- [Background] Rocha-Singh KJ, Zeller T, Jaff MR. Peripheral arterial calcification: prevalence, mechanism, detection, and clinical implications. Catheter Cardiovasc Interv. 2014 May 1;83(6):E212-20. doi: 10.1002/ccd.25387. Epub 2014 Feb 10. PMID 24402839

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT06416644/Prot_SAP_000.pdf